CLINICAL TRIAL: NCT03988244
Title: Clinical Study of the HeartLight X3 Endoscopic Ablation System (EAS) With Excalibur Balloon Compared to HeartLight System in the Treatment of Symptomatic Persistent Atrial Fibrillation
Brief Title: HeartLight X3 Endoscopic Ablation System With Excalibur Balloon for Treatment of Symptomatic Persistent AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-4911
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HeartLight X3 (Experimental): Pulmonary vein isolation using HeartLight X3
  Interventions: Device: HeartLight X3

INTERVENTIONS:
Device: HeartLight X3 — Pulmonary vein isolation

SUMMARY:
The objective of the study is to demonstrate the improved ablation and procedure times of the HeartLight X3 compared to the original HeartLight catheter in the treatment of persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* early persistent AF, failure of at least one AAD, others

Exclusion Criteria:

* overall good health as established by multiple criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Ablation time | Acute - at the end of the index procedure
  Ablation time

SECONDARY OUTCOMES:
Procedure time | Acute - at the end of the index procedure
  Procedure time
PV Isolation | Acute - at the end of the index procedure
  Percent of isolated pulmonary veins
PAE Rate | 30 Days
  Primary Adverse Event rate
AF Free Rate | 6 and 12 months
  6- and 12-month chronic results

CONTACTS AND LOCATIONS:
Overall Officials: Burke T. Barrett, Study Director — CardioFocus, Inc.
Locations (1):
- Nemocnice Na Homolce, Prague, Czechia